CLINICAL TRIAL: NCT06481852
Title: A Placebo-controlled, Randomized Clinical Trial to Assess the Safety, Feasibility, and Pharmacokinetics of Microbiota Transplant Therapy With Antibiotic Preconditioning and Fiber Supplementation in Patients With Pulmonary Arterial Hypertension
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CV-2024-32994
Record Dates: First submitted 2024-06-24; First posted 2024-07-01 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — monooxyethylene trimethylolpropane tristearate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Drug group (Experimental): PAH patients randomized to MTT with antibiotic preconditioning + fiber supplementation
  Interventions: Drug: MTT with antibiotic preconditioning + fiber supplementation
- Control 1 (Active Comparator): MTT with antibiotic preconditioning + placebo supplementation
  Interventions: Drug: MTT with antibiotic preconditioning + placebo supplementation
- Control 2 (Placebo Comparator): placebo + placebo supplementation.
  Interventions: Other: MTT with placebo + placebo supplementation.

INTERVENTIONS:
Drug: MTT with antibiotic preconditioning + fiber supplementation — MTT will in a capsule form composed of freeze-dried, encapsulated intestinal microbiota from healthy donors. Fiber supplementation will be 10-14 gm oral fiber supplement. Patients will be followed at week 1, week 2, week 4, week 12, and week 24. Patient will undergo stool sample collection at baseline, week 1, week 4, and week 12, blood sample collection at baseline, week 4, and week, 12. In addition, patient will undergo an echocardiogram, six-minute walk test (6MWT) and quality of life questionnaire at baseline and at week 12.
  Arms: Drug group
Drug: MTT with antibiotic preconditioning + placebo supplementation — MTT will in a capsule form composed of freeze-dried, encapsulated intestinal microbiota from healthy donors. Patients will be followed at week 1, week 2, week 4, week 12, and week 24. Patient will undergo stool sample collection at baseline, week 1, week 4, and week 12, blood sample collection at baseline, week 4, and week, 12. In addition, patient will undergo an echocardiogram, six-minute walk test (6MWT) and quality of life questionnaire at baseline and at week 12.
  Arms: Control 1
Other: MTT with placebo + placebo supplementation. — MTT will in a capsule form composed of freeze-dried, encapsulated intestinal microbiota from healthy donors. Patients will be followed at week 1, week 2, week 4, week 12, and week 24. Patient will undergo stool sample collection at baseline, week 1, week 4, and week 12, blood sample collection at baseline, week 4, and week, 12. In addition, patient will undergo an echocardiogram, six-minute walk test (6MWT) and quality of life questionnaire at baseline and at week 12.
  Arms: Control 2

SUMMARY:
This pilot clinical trial will evaluate the initial safety, feasibility, and pharmacokinetics of microbiota transplant therapy (MTT) with antibiotic pre-conditioning and fiber supplementation vs. placebo in patients with pulmonary arterial hypertension (PAH). This trial will inform development of future trials of MTT as a treatment for PAH. 24 PAH patients will be randomized to receive either MTT with antibiotic preconditioning + fiber supplementation, MTT with antibiotic preconditioning + placebo supplementation, or placebo + placebo supplementation. MTT will in a capsule form composed of freeze-dried, encapsulated intestinal microbiota from healthy donors. Fiber supplementation will be 10-14 gm oral fiber supplement. Patients will be followed at week 1, week 2, week 4, week 12, and week 24. Patient will undergo stool sample collection at baseline, week 1, week 4, and week 12, blood sample collection at baseline, week 4, and week,12. In addition, patient will undergo an echocardiogram, six-minute walk test (6MWT) and quality of life questionnaire at baseline and at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated consent form
* Ages 18-75
* Diagnosis of PAH
* On stable treatment for PAH for one month prior to enrollment
* Able to swallow capsules
* Able to provide blood sample and fecal sample
* Stated willingness to comply with all study procedures and availability for the duration of trial to follow-up by telephone, in-person, email, and/or video visits or correspondence.

Exclusion Criteria:

* Dysphagia to pills
* Clinically active inflammatory bowel disease
* Pregnancy or breastfeeding. A pregnancy test will be obtained from females of child- bearing potential at the screening visit or day 1 (prior to the receipt of MTT). Patients with a positive pregnancy test will be excluded. A negative result will be required for subjects who are females of child-bearing potential to receive MTT. Patients will be counseled to avoid pregnancy which is the standard of care for patients with PAH.
* Life expectancy of < 6 months
* Presence of ileostomy or colostomy
* Patients on immunosuppressants (calcineurin inhibitors, prednisone ≥ 20 mg/day, methotrexate, azathioprine, immunosuppressive biologics, JAK inhibitors).
* Patients with neutropenia (an absolute neutrophil count < 0.5 x 10 9 cells/L) obtained on a complete blood count with differential at screening
* History of solid organ or bone marrow transplant
* Anticipated recurrent antibiotic use (patients with frequent urinary tract infections or sinusitis)
* History of severe anaphylactic food allergy
* History of celiac disease
* Patients receiving cancer chemotherapy, immunotherapy, or radiation
* Patients with severe Irritable bowel syndrome (IBS) defined by an IBS score >250

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
donor engraftment comparison | week 12
  The difference in donor microbiota engraftment between the three study groups at week 12

SECONDARY OUTCOMES:
safety of MTT with antibiotic preconditioning and fiber supplementation in patients with PAH | week 12
  The difference in frequency of serious adverse events and other adverse events between the three study groups
feasibility of MTT with antibiotic preconditioning and fiber supplementation in patients with PAH | week 12
  The differences in proportion of subjects taking 100% of the MTT per protocol between the three study groups
change in inflammatory markers | week 12
  The differences in the change in circulating markers of inflammation and microbial metabolites from baseline to week 12 between the three study groups
compare right ventricular function, measure 1 | week 12
  The differences in the change in six-minute walk distance (6MWD) from baseline to week 12 between the three study groups
compare right ventricular function | week 12
  The differences in the change in right ventricular ejection fraction from baseline to week 12 between the three study groups
compare right ventricular function | week 12
  The differences in the change in quality of life survey from baseline to week 12 between the three study groups

CONTACTS AND LOCATIONS:
Overall Officials: Thenappan Thenappan, MD, Principal Investigator — University of Minnesota; Levi Teigen, MD, PhD, Principal Investigator — University of Minnesota; Alexander Khoruts, MD, Principal Investigator — University of Minnesota; Christopher Staley, PhD, Principal Investigator — University of Minnesota; Kurt Prins, MD,PhD, Principal Investigator — University of Minnesota; Edward Weirs, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No